CLINICAL TRIAL: NCT02463929
Title: Dyphenhidramine Effect on Prevention of Sevoflurane Induced Post Anesthesia Agitation in Pediatric
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitas Diponegoro (Other)
Collaborators: Permata Sari Hospital for Plastic Surgery (Unknown)
Responsible Party: Principal Investigator, Ika Cahyo Purnomo, Doctor, Universitas Diponegoro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UDiponegoro
Record Dates: First submitted 2015-05-18; First posted 2015-06-04 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Specified Sedative; Hypnotic
Keywords: Diphenhydramine; emergence agitation; pediatric anesthesia; PAEDS; Withdrawal
MeSH Terms: conditions — Emergence Delirium | interventions — Diphenhydramine; Saline Solution; Ketamine; Sevoflurane; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- diphenhydramine (Experimental): Subject sedated with sevoflurane, and given bilateral extraoral infraorbital block with 0,125% bupivacaine. Subject injected 0,5mg/kg diphenhydramine intravenously, 15 minutes prior to discontinuation of sevoflurane. If subject develop agitation, 0,1 mg/kg ketamine is administered
  Interventions: Drug: Diphenhydramine; Drug: Ketamine; Drug: Sevoflurane; Drug: Bupivacaine
- control (Placebo Comparator): Subject sedated with sevoflurane, and given bilateral extraoral infraorbital block with 0,125% bupivacaine. Subject injected 0,5cc/kg normal saline intravenously, 15 minutes prior to discontinuation of sevoflurane. If subject develop agitation, 0,1 mg/kg ketamine is administered
  Interventions: Drug: normal saline; Drug: Ketamine; Drug: Sevoflurane; Drug: Bupivacaine

INTERVENTIONS:
Drug: Diphenhydramine — Intravenous Injection
  Arms: diphenhydramine
Drug: normal saline — Intravenous Injection
  Other Names: NaCl 0,9%
  Arms: control
Drug: Ketamine — Ketamine 0,1 mg/kg intravenously used as rescue tranquilizer if the subject becomes agitated, repeated dose of 0,05 mg/kg every minute can be given if the agitation does not resolve, maximum ketamine dose for tranquilizer 0,25 mg/kg to prevent deep sedation
Drug: Sevoflurane — Sevoflurane as single sedation agent for general anesthesia in both arm. 8% Sevoflurane in 100% oxygen used as induction agent, and 2% sevoflurane in 50% oxygen used as maintenance agent
Drug: Bupivacaine — Bilateral extraoral infraorbital nerve block with 0,125% Bupivacaine as analgetic for operation and post operation.

SUMMARY:
The purpose of this study is to investigate the effect of diphenhydramine on the prevention of sevoflurane induced emergence delirium/ agitation in pediatrics. The Investigators hypothesis is that it reduce the incidence of sevoflurane induced emergence delirium/ agitation.

DETAILED DESCRIPTION:
This is an experimental clinical trial in double-blinded randomized controlled design on 50 children aged 10 months to 21 months who underwent general anesthesia with sevoflurane for labioplasty surgery. Fifteen minutes before inhalation anesthetics were discontinued, the subjects were randomly given a placebo or a single dose of diphenhydramine 0, 5 mg / kg intravenously. Subjects were extubated and observed in the recovered space conscious for any agitation or emergence delirium and feasability to return to the ward. Agitation or emergence delirium was assessed by the Pediatric Emergence Agitation and Delirium Score (PAEDS) whereas feasability to return to the ward scored with the Steward score. When PAEDS> 10 patients were assessed to be agitated or having emergence delirium and administeres rescue tranquilizer ketamine 0.1 mg / kg. Total rescue tranquilizers and clinically significant adverse effects of drugs also recorded.

ELIGIBILITY:
Inclusion Criteria:

ASA I or 2

* no cardiovascular, respiratory or neurologic congenital anomalies
* no allergic reactions, or any contraindication to drugs used in this trial ever documented

Exclusion Criteria:

* congenital anomalies recognized/diagnosed during trial procedures
* hemmorhage > 15% EBV
* shock or other major anesthesia or surgical complications during trial procedures (hipoxia, atelectasis, unintended disconection of ETT or IV line)

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Incidence of sevoflurane induced post anesthesia agitation | 10 minutes post extubation

SECONDARY OUTCOMES:
Amount of rescue Ketamine used | 1 minute post extubation, at emergence, 15 minute post extubation
  Administration of 0,1 mg/kg ketamine intravenously if the patient gets agitated
Significant adverse events | 1 minute post extubation, at emergence, 15 minute post extubation
  Any respiratory or cardiovascular events during observation in recovery room
Mean Pediatric Emergence Agitation and Delirium Score (PAEDS) | 1 minute post extubation
Mean Pediatric Emergence Agitation and Delirium Score (PAEDS) | at emergence
Mean Pediatric Emergence Agitation and Delirium Score (PAEDS) | 15 minute post extubation
Incidence of sevoflurane induced post anesthesia agitation | 1 minute post extubation
Incidence of sevoflurane induced post anesthesia agitation | 15 minute post extubation
Length of stay in recovery room | up to 15 minutes post extubation

CONTACTS AND LOCATIONS:
Overall Officials: Johan Mr Arifin, dr, Study Director — Universitas Diponegoro

REFERENCES:
- [Background] Varughese AM, Rampersad SE, Whitney GM, Flick RP, Anton B, Heitmiller ES. Quality and safety in pediatric anesthesia. Anesth Analg. 2013 Dec;117(6):1408-18. doi: 10.1213/ANE.0b013e318294fb4a. PMID 24257392
- [Background] Cohen IT, Finkel JC, Hannallah RS, Hummer KA, Patel KM. The effect of fentanyl on the emergence characteristics after desflurane or sevoflurane anesthesia in children. Anesth Analg. 2002 May;94(5):1178-81, table of contents. doi: 10.1097/00000539-200205000-00023. PMID 11973185
- [Background] Koner O, Ture H, Mercan A, Menda F, Sozubir S. Effects of hydroxyzine-midazolam premedication on sevoflurane-induced paediatric emergence agitation: a prospective randomised clinical trial. Eur J Anaesthesiol. 2011 Sep;28(9):640-5. doi: 10.1097/EJA.0b013e328344db1a. PMID 21822077
- [Background] Abdallah C, Hannallah R. Premedication of the child undergoing surgery. Middle East J Anaesthesiol. 2011 Jun;21(2):165-74. No abstract available. PMID 22435268
- [Background] Aouad MT, Nasr VG. Emergence agitation in children: an update. Curr Opin Anaesthesiol. 2005 Dec;18(6):614-9. doi: 10.1097/01.aco.0000188420.84763.35. PMID 16534301
- [Background] Simons FE, Simons KJ. Clinical pharmacology of H1-antihistamines. Clin Allergy Immunol. 2002;17:141-78. No abstract available. PMID 12113216